CLINICAL TRIAL: NCT03161522
Title: A Randomized Trial Comparing Early Local Chemoradiation Therapy +/- Surgery Versus Systemic Therapy for Patients With Esophageal or Gastric Cancer With Oligometastases
Brief Title: Chemotherapy With or Without Radiation or Surgery in Treating Participants With Oligometastatic Esophageal or Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0972; NCI-2018-01202 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0972 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Gastric Adenocarcinoma; Oligometastasis; Stage IV Esophageal Adenocarcinoma AJCC v7; Stage IV Esophageal Cancer AJCC v7; Stage IV Gastric Cancer AJCC v7
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms; Stomach Neoplasms | interventions — Capecitabine; Drug Therapy; Fluorouracil; dehydroftorafur; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (maintenance chemotherapy) (Experimental): Participants receive fluorouracil and capecitabine per instructions of the treating physician in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capecitabine; Drug: Chemotherapy; Drug: Fluorouracil
- Group II (local therapy) (Experimental): Participants receive fluorouracil and capecitabine and undergo RT per instructions of the treating physician in the absence of disease progression or unacceptable toxicity. Participants may also undergo surgery to some or all of the remaining sites of disease as is clinically prudent and indicated by treating physician.
  Interventions: Drug: Capecitabine; Drug: Chemotherapy; Procedure: Conventional Surgery; Drug: Fluorouracil; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Capecitabine — Patients will receive 5-fluorouracil (5-FU) and capecitabine as maintenance chemotherapy.
  Other Names: Ro 09-1978/000; Xeloda
Drug: Chemotherapy — Receive induction chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Procedure: Conventional Surgery — Undergo surgery
  Arms: Group II (local therapy)
Drug: Fluorouracil — Patients will receive 5-fluorouracil (5-FU) and capecitabine as maintenance chemotherapy.
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
  Arms: Group II (local therapy)

SUMMARY:
This phase II trial studies how well chemotherapy with or without radiation or surgery works in treating participants with esophageal or gastric cancer that has spread to less than 3 places in the body (oligometastatic). Drugs used in chemotherapy, such as fluorouracil and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Surgery, such as complete surgical resection, may stop the spread of tumor cells by surgically removing organs or tumors. Giving chemotherapy with radiation or surgery may work better than chemotherapy alone in treating participants with oligometastatic esophageal or gastric cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether esophageal or gastric patients with oligometastatic cancer without disease progression after first line chemotherapy therapy will demonstrate improved overall survival (OS) with early local therapy (concurrent chemotherapy/radiation and surgery).

SECONDARY OBJECTIVES:

I. Assess the relationships between progression-free survival and overall survival between both treatment arms.

II. Report local control, loco-regional control. III. Report time to progression of distant metastases. IV. Report toxicity.

OUTLINE:

Participants receive induction chemotherapy for a minimum of 6 cycles and a maximum of 8 cycles in the absence of disease progression or unacceptable toxicity. Participants are then randomized to 1 of 2 groups.

GROUP I (MAINTENANCE CHEMOTHERAPY): Participants receive fluorouracil and capecitabine per instructions of the treating physician in the absence of disease progression or unacceptable toxicity.

GROUP II (LOCAL THERAPY): Participants receive fluorouracil and capecitabine and undergo radiation therapy (RT) per instructions of the treating physician in the absence of disease progression or unacceptable toxicity. Participants may also undergo surgery to some or all of the remaining sites of disease as is clinically prudent and indicated by treating physician.

After completion of study treatment, participants are followed up at 4-8 weeks, 2-3 months, every 3-6 months for up to 3 years, and then every 6-12 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a pathologic diagnosis of tumor biopsy or FNA of esophageal or gastric cancer of adenocarcinoma histology
* The patient is staged with EGD and PET/CT scan.
* The patient has three or less observable metastatic lesions. Patients may have three or less radiographically visible metastatic lesions at diagnosis or if have regressed to three or less metastatic lesions after induction chemotherapy at time of randomization. The patient must have pathologic confirmation and or radiologically visible disease. For esophageal tumors, the maximal dimension of the primary tumor may not provide reproducible measurements for RECIST and may not be visible on CT or PET/CT at diagnosis or after induction chemotherapy. Accordingly, patients are eligible regardless of the imaging measurements of the primary tumor. Additionally, in patients with non-measurable metastases, patients are eligible if there is pathology confirming metastases from a distant site. However, biopsy of a metastatic site is not required if there are visible metastases on imaging (such as ultrasound, diagnostic CT , EUS, PET/CT).

  * The patient has three or less observable metastatic lesions by diagnostic scans (CT scan, PET/CT, eEndoscopic ultrasound, MRI, or bone scan). Metastatic lesions include distant M1 lymph node group; which will be counted as one site (M1 metastatic lymph nodes to include cervical, mediastinal, gastric, retroperitoneal lymph nodes will be counted as one lesion).
  * Osseous metastases or visceral metastases will each count as one metastatic site.
  * Each CNS metastases will count as one metastatic site.
  * Satellite lesions in the primary esophageal malignancy such as skipped esophageal primaries are not considered metastatic sites. Symptomatic metastatic sites can be treated locally prior to randomization or by palliative radiation.
  * Symptomatic metastatic sites may be treated with radiation or surgery prior to enrollment.
* Patient ECOG of 0-2, with life expectancy of at least 6 months
* Patients age >18 yrs old but <80 yrs old and signed informed consent
* Women of child-bearing age must have pregnancy test at time of enrollment, agree to use of adequate contraception (birth control hormone or barrier method) for the duration of the study and for six months after discontinuation of systemic agents.

Exclusion Criteria:

* Patients with prior chemotherapy or radiation therapy for their diagnosis of esophageal or gastric cancer. Patients with prior radiation therapy to same site for another diagnosis of cancer. Note: Patients may receive palliative radiation to their symptomatic sites of metastases but not definitive local therapy to esophageal or gastric primary prior to randomization. All patients may be enrolled on protocol then start systemic therapy; if they do not have evidence of disease progression at re-staging following initial therapy, they may be randomized.
* Patients with fistula documented radiographically or by EDG/EUS, EBUS.
* Patients with life expectancy less than 6 months, ECOG >3
* Female patients who are pregnant confirmed by bHCG lab test.
* Patient has history of uncontrolled angina, congestive heart failure or recent MI within 6 months.
* Nursing females
* Patients in poor nutritional state
* Patients with:

  * Severely depressed bone marrow function
  * Potentially serious infections
  * Known hypersensitivity to 5-fluorouracil
  * Known or suspected to have a dihydropyrimidine dehydrogenase deficiency (as these patients are at a greater risk of experiencing symptoms of toxicity)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 6 years
  OS distributions in the two arms will be estimated by the method of Kaplan and Meier. Bayesian piecewise exponential regression will be used to assess the relationships between each of OS and PFS, and patients' covariates and treatment arm.

SECONDARY OUTCOMES:
Local progression-free survival (PFS) | Up to 6 years
  PFS distributions in the two arms will be estimated by the method of Kaplan and Meier. Bayesian piecewise exponential regression will be used to assess the relationships between each of OS and PFS, and patients' covariates and treatment arm.
Distant PFS | Up to 6 years
  PFS distributions in the two arms will be estimated by the method of Kaplan and Meier. Bayesian piecewise exponential regression will be used to assess the relationships between each of OS and PFS, and patients' covariates and treatment arm.
Incidence of adverse events | Up to 6 years
  Graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time to local or regional disease recurrence | Up to 6 years
  To be analyzed by Bayesian piecewise regression to assess their relationships with treatment arm and prognostic covariates.

OTHER OUTCOMES:
Time to local disease recurrence | Up to 6 years
  To be analyzed by Bayesian piecewise regression to assess their relationships with treatment arm and prognostic covariates.
Time to disease progression | Up to 6 years
  To be analyzed by Bayesian piecewise regression to assess their relationships with treatment arm and prognostic covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Nhu Nguyen, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org